CLINICAL TRIAL: NCT06620653
Title: Heart Failure Virtual Ward Research Study
Acronym: HF-VW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Derek O'Keeffe, Principal Investigator, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Heart Failure Virtual Ward
Record Dates: First submitted 2024-07-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. half of the participants will be in the tele monitoring group while the other half will be in the current standard of care group
Masking Description: the participants will be randomised using REDCAP software but there will be no masking performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Active Comparator): All patients with a recent admission for decompensated heart failure are seen in a first face-to-face appointment within two weeks of discharge as per current 2021 ESC Heart Failure Guidelines.
  The standard care group will receive the usual nurse lead structured follow up and patients in the usual care will have a face-to-face appointment at week 6 and 12, and all the other contacts will be phone calls or face-to-face
  Interventions: Other: Standard Care
- Telemonitoring (Experimental): After the initial face-to-face appointment the telemonitoring group will have appointments at week 4 (phone call or videoconference), week 6 (videoconference), week 8 (phone call or videoconference) and week 12 (videoconference). In total, the patients will have 6 structured appointments.
  Extra phone calls, videoconferences, and face-to-face visits will be made at any time, depending on the patient's needs, irrespective of the assigned group.
  Patients assigned to the intervention group will receive a tablet (if the patients do not have a tablet, computer or smartphone), a weight scale and a blood pressure monitor. The patients will provide daily biometric data (weight, heart rate and blood pressure) and report symptoms through four questions to capture worsening symptoms of the cardiac condition.
  The system will generate warning alarms (biometrics out of range or symptom reporting) and alerts (information related to the function of the household devices).
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — Patients assigned to the intervention group will receive a tablet (if the patients do not have a tablet, computer or smartphone), a weight scale and a blood pressure monitor. The patients will provide daily biometric data (weight, heart rate and blood pressure) and report symptoms through four questions to capture worsening symptoms of the cardiac condition.
  Arms: Telemonitoring
Other: Standard Care — patients with a recent admission for heart failureare seen in a first face-to-face appointment within two weeks of discharge as per current 2021 ESC Heart Failure Guidelines with face-to-face follow up at 6 and 12 weeks.
  Arms: Standard Care

SUMMARY:
The main aim will be to evaluate whether a follow-up with virtual wards reduces HF hospitalisation at three months follow-up. Hospital admission will be defined as any hospital admission, or an emergency room stay of more than 24 h requiring IV diuretics.

The secondary objectives will be to evaluate whether this intervention reduces all-cause mortality, all-cause hospitalisation at three months, is cost-effectiveness, is associated with a higher percentage of prescription and dose of prognostic medication and improves the quality of life. To assess the potential long-term effects of the virtual wards follow-up, we will evaluate whether this intervention reduces all-cause mortality and HF hospitalisation at 6- and 12-months by a telephone call/virtual outpatients' appointment.

The study outcomes will be ascertained at each visit. Given the study design, it is impossible to assess the endpoints in a blinded manner. Clinical events during the study will be adjudicated by an operational committee whose members will be unaware of the group assignment.

DETAILED DESCRIPTION:
This is a randomized, controlled, multicentre, parallel-group trial in which we will consecutively include all patients over 18 years of age with a recent hospitalisation due to decompensated HF and randomise them to usual care vs. telemedicine follow-up. Any stay in the emergency department or ward for over 24 hours that required treatment with intravenous diuretic will be considered an hospitalisation.

The heart failure diagnosis will be made according to the 2021 ESC Heart Failure Guidelines.

The study will be registered at ClinicalTrials.gov. The study will be guided by good clinical practice (GCP), in accordance with the Declaration of Helsinki and the laws and regulations applicable in Ireland. Written approval from the appropriate Ethics Committees will be required, and each patient will provide written informed consent before enrolling in the study.

Patients will be recruited from the participant hospitals (Portiuncula University Hospital and Galway University Hospital).

Inclusion criteria: The study will include adult patients (≥ 18 years) with a recent hospitalisation. We will include all ranges of ejection fraction, and also patients with known and de novo heart failure.

The main exclusion criteria will be:

* Patients who decline to participate in the study.
* Patient in palliative care or with a life expectancy of less than one year.
* Patients referred to skilled nursing facilities or nursing homes at hospital discharge.
* Patients with planned intervention on the mitral or aortic valve during admission or scheduled early after discharge.
* Planned haemodialysis.
* Patients included in other randomized controlled trials.
* Patients who, at the investigator's discretion, are considered unable to participate in the study, mainly due to a previous history of non-compliance with medication and follow-up appointments, language barrier, or moderate or severe cognitive impairment without the support of a family member/caregiver.
* Patients with asymptomatic (NYHA class I) left ventricular dysfunction, usually in the setting of an acute myocardial infarction.

The lack of information technology (IT) literacy will not be an exclusion criterion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with a recent hospitalisation.
* Known ejection fraction and NYHA Class
* Known or de novo Heart Failure
* Patient or carer able to speak and understand English/Irish
* Willing to participate in the study.
* Within catchment area of the Saolta group.

Exclusion Criteria:

* Patients who decline to participate in the study.
* Patient in palliative care or with a life expectancy of less than one year.
* Patients referred to skilled nursing facilities or nursing homes at hospital discharge.
* Patients with planned intervention on the mitral or aortic valve during admission or scheduled early after discharge.
* Planned haemodialysis.
* Patients included in other randomized controlled trials.
* Patients who, at the investigator's discretion, are considered unable to participate in the study, mainly due to a previous history of non- compliance with medication and follow-up appointments, language barrier, or moderate or severe cognitive impairment without the support of a family member/caregiver.
* Patients with asymptomatic (NYHA class I) left ventricular dysfunction, usually in the setting of an acute myocardial infarction.
* The lack of information technology (IT) literacy will not be an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in re-admission rates | three months
  Whether a follow-up with virtual wards reduces HF hospitalisation at three whether a follow up with virtual wards reduces HF hospitalisation at three months follow-up

SECONDARY OUTCOMES:
All cause mortality | 12 months
  Whether HF virtual wards reduces all cause mortality
Financial Cost of virtual ward in comparison to the standard care | 3 months
  Analysis of the financial implications of using the virtual heart failure ward in comparison to the cost of standard heart failure care

CONTACTS AND LOCATIONS:
Overall Officials: Derek O&amp;#39;Keeffe, MD, PhD, Principal Investigator — Galway University Hospitals/University of Galway
Locations (1):
- Portiuncula University Hospital, Ballinasloe, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller-Davis C, Marden S, Leidy NK. The New York Heart Association Classes and functional status: what are we really measuring? Heart Lung. 2006 Jul-Aug;35(4):217-24. doi: 10.1016/j.hrtlng.2006.01.003. PMID 16863893